CLINICAL TRIAL: NCT01348906
Title: Effect of Intermittent Normoxic Cardiopulmonary Bypass on Myocardial Reperfusion Injury in Adult Valve Replacement
Brief Title: Intermittent Normoxia Reduces Myocardial Reperfusion Injury
Acronym: INCPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Shengxi Chen, Department of Cardiothoracic Surgery, Xiangya Hospital, Central South University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCPB
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Hyperoxia
Keywords: cardiopulmonary bypass
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermittent normoxia (Experimental): Repeated brief normoxic reperfusion during cardioplegia arrest in adult valve replacement
  Interventions: Procedure: intermittent normoxia

INTERVENTIONS:
Procedure: intermittent normoxia — 3 cycles of 5/5 min normoxia/hyperoxic reperfusion during cardioplegia arrest in adult valve replacement

SUMMARY:
This study aims to determine the effect of intermittent normoxic cardiopulmonary bypass (CPB) on inflammatory response, oxidative stress and myocardial reperfusion injury in adult patients undergoing valve replacement. The investigators hypothesized that nuclear factor kappa B (NFkB) was involved in regulating gene expression of myocardial inflammatory factor.

DETAILED DESCRIPTION:
Methods:Patients meeting the requirement will be randomized into 2 groups: the control group received hyperoxic reperfusion (PaO2 180-250 mmHg) throughout CPB as routine; the treatment group underwent 3 cycles of 5/5 min normal/high oxygenation (PaO2 80-150/180-250 mmHg) during cardioplegia arrest, and maintained the same hyperoxia as the control group in the rest time of CPB. The clinical data of inotropes requirement, drainage, ventilation and intensive care time will be recorded. Venous blood samples will be taken perioperatively for detecting concentration of troponin I (cTnI), tumor necrosis factor-α , interleukin-6, 10, and malondialdehyde (MDA). Atrial biopsies will be removed before cardioplegia arrest and 30min after aortic de-clamping to determine the extent of neutrophil infiltration (myeloperoxidase activity), NFkB binding DNA activity, and gene expression of inflammatory factors (TNF-α, IL-6, 10).

Statistical analysis:A sample size of at least 32 patients in each group was needed to have a power of 90%, significance at the two-side 5% level, on the basis that a SD of 0.2 ng/ml and a difference in peak serum cTnI release of about 0.15 ng/ml between control and conditioned patients was determined.

Expected Results: The treatment group will have significantly lower release of cTnI, inflammatory factors, and MDA during CPB and afterwards. Intermittent normoxia may be related to less myocardial inflammation characterized by decreased myeloperoxidase activity, gene expression of inflammatory factors, the later may result from reduced activity of NFkB binding to DNA after reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* rheumatic heart valve disease requiring selective aortic or double valve(aortic and mitral valve) replacement

Exclusion Criteria:

* infective endocarditis congenital valve disease previous cardiac surgery complicated with diabetes, coronary artery disease, hypertension or peripheral vascular disease.

receiving aspirin, corticosteroids, angiotensin-converting enzyme inhibitors or statin perioperatively

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
plasma concentration of troponin I | within the first 24h after cardiac surgery

SECONDARY OUTCOMES:
gene expression of TNFa, IL-6, and IL-10 in myocardium | 30 min after aotic de-clamping

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery, Xiangya Hospital, Central South University, Changsha, Hunan, China